CLINICAL TRIAL: NCT06625996
Title: Examining the Effectiveness of Carbohydrate Loading as a Nursing Intervention in Enhanced Recovery After Surgery: A Comprehensive Analysis of Protocol Compliance and Patient Outcomes
Brief Title: Examining the Effectiveness of Carbohydrate Loading as a Nursing Intervention in Enhanced Recovery After Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAK Medical and Health Sciences University (Other)
Responsible Party: Principal Investigator, Mona Gamal, Assistant Professor, RAK Medical and Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3380031
Record Dates: First submitted 2024-09-30; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Diet, Carbohydrate Loading

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental)
  Interventions: Dietary Supplement: carbohydrate loading
- control (Placebo Comparator): No intervention
  Interventions: Dietary Supplement: carbohydrate loading

INTERVENTIONS:
Dietary Supplement: carbohydrate loading — Preoperative carbohydrate loading

SUMMARY:
The concept of Enhanced Recovery After Surgery (ERAS) protocols has revolutionized perioperative care by promoting a series of evidence-based practices aimed at reducing surgical stress and improving patient outcomes. Among these practices, preoperative carbohydrate loading has emerged as a significant intervention designed to mitigate the adverse metabolic effects of surgery

ELIGIBILITY:
Inclusion Criteria:

- Cardiovascular disease

Exclusion Criteria:

Insulin dependent diabetes

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-11-06 (Estimated); Study Completion 2026-10-06 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay post cardio thoracic surgery | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No